CLINICAL TRIAL: NCT06955585
Title: Efficacy of Lipid-containing Artificial Tears in the Treatment of Dry Eye
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Danijel Mikulic, MD, University Hospital Sestre Milosrdnice
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DED-2025
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Dry Eye Disease; Dry Eye; Dry Eye, Evaporative
Keywords: dry eye; artificial tears
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proluxx Treatment Group (Experimental): Group that will use topical artificial tear spray applied to closed eyelids four times daily for 28 days.
  Interventions: Device: Proluxx Artificial Tear Spray

INTERVENTIONS:
Device: Proluxx Artificial Tear Spray — Topical artificial tear spray applied to closed eyelids four times daily for 28 days.
  Other Names: Proluxx Duo sprej za oko

SUMMARY:
This clinical study involves patients with Dry Eye Disease (DED) who are visiting an ophthalmology outpatient clinic. Eligible participants must have an Ocular Surface Disease Index (OSDI) score ≥14 and <50, and at least one positive diagnostic test: tear break-up time (TBUT) <7 seconds, Schirmer I test <10 mm/5 min, or positive corneal staining based on the Oxford grading scale. At baseline, tear film thickness will be measured using Pentacam imaging. Participants will then receive Proluxx eye spray, applied four times daily for 28 days. After this treatment period, a follow-up examination with all baseline assessments will be repeated.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the effects of Proluxx artificial tear spray in patients diagnosed with Dry Eye Disease (DED). Participants are recruited from an ophthalmology outpatient clinic and must have had symptoms of DED for at least 3 months. Inclusion criteria include an Ocular Surface Disease Index (OSDI) score between 14 and 50 and at least one positive diagnostic test: tear break-up time (TBUT) <7 seconds, Schirmer I test (≤10 mm/5 min), or positive corneal staining based on the Oxford grading scheme. In addition, participants must not have used artificial tears for at least two weeks prior to enrollment, even if they were previously on such therapy.

Exclusion criteria include the use of systemic or topical corticosteroids, active ocular infection, or ocular surgery within the last 3 months.

The goal of the study is to classify patients based on DED subtype: hyposecretory, evaporative, or mixed. The study will analyze clinical parameters at baseline, including OSDI score, TBUT, Schirmer test, Oxford staining, CPTFT (central precorneal tear film thickness) measured by Pentacam, BCVA (best corrected visual acuity), intraocular pressure (IOP), and risk factors. Participants will use Proluxx artificial tear spray four times daily for 28 days. After the treatment period, all baseline assessments will be repeated.

The study will compare clinical findings from Day 0 and Day 28 to assess changes in ocular surface health and tear film quality following therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ocular Surface Disease Index (OSDI) score between 14 and 50 and at least one positive diagnostic test: tear break-up time (TBUT) <7 seconds, Schirmer I test (≤10 mm/5 min), or positive corneal staining based on the Oxford grading scheme. In addition, participants must not have used artificial tears for at least two weeks prior to enrollment, even if they were previously on such therapy

Exclusion Criteria:

* use of systemic or topical corticosteroids, active ocular infection, or ocular surgery within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in Central Precorneal Tear Film Thickness (CPTFT) | Baseline (Day 0) and Day 28
  Change in central precorneal tear film thickness measured using Pentacam imaging between baseline and after 28 days of treatment with Proluxx artificial tear spray.
Change in Ocular Surface Disease Index (OSDI) Score | Baseline and Day 28
  Change in OSDI questionnaire score to evaluate improvement in symptoms of dry eye disease after 28 days of therapy.

SECONDARY OUTCOMES:
Change in Tear Break-Up Time (TBUT) | Baseline and Day 28
  Measurement of tear film stability by TBUT test, comparing values at baseline and after 28 days of treatment.
Change in Corneal Staining Grade (Oxford Scale) | Baseline and Day 28
  Assessment of ocular surface damage using Oxford grading of corneal staining at baseline and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ivanka Petric Vicković, Prof,MD,PHD, Study Director — Eye Department of UHC Sestre milosrdnice Zagreb
Locations (1):
- UHC Sestre milosrdnice, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No